CLINICAL TRIAL: NCT02711683
Title: DL-3-n-butylphthalide Treatment in Patients With Mild to Moderate Alzheimer's Disease Already Receiving Donepezil : A Multi Center, Prospective Cohort Stud
Brief Title: DL-3-n-butylphthalide Treatment in Patients With Mild to Moderate Alzheimer's Disease Already Receiving Donepezil
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2015-027
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-n-butylphthalide; Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DL-3-n-butylphthalide group: using DL-3-n-butylphthalide treatment in patients with mild to moderate AD already receiving donepezil
  Interventions: Drug: DL-3-n-butylphthalide; Drug: Donepezil
- donepezil group: only using donepezil treatment in patients with mild to moderate AD
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: DL-3-n-butylphthalide — the patients with mild to moderate AD have already been prescribed the drugs,we just observed passively.
  Other Names: NBP
  Groups: DL-3-n-butylphthalide group
Drug: Donepezil — the patients with mild to moderate AD have already been prescribed the drugs,we just observed passively.
  Other Names: Aricept

SUMMARY:
Alzheimer's disease (AD) is the commonest cause of dementia. There is no effective treatment to cure the disease. Cholinesterase inhibitors, such as donepezil, are widely recommended to patients with mild to moderate AD. But the cognitive function of most of the patients using donepezil gradually aggravate, with Mini-Mental State Examination(MMSE) score falling by 2 points per year on average, and donepezil cannot effectively delay AD progress.

DL-3-n-butylphthalide(NBP) is a synthetic chiral compound containing L- and D-isomers of butylphthalide. It is developed from L-3-n-butylphthalide, which was initially isolated as a pure component from seeds of Apium graveolens in 1978 by researchers of Institute of Medicine of Chinese Academy of Medical Sciences. Studies in the past several decades have demonstrated that NBP is effective in alleviating oxidative damage and mitochondria dysfunction, improving microcirculation. NBP was approved by the State Food and Drug Administration of China (SFDA) as a therapeutic drug for treatment of ischemic stroke in 2005 Not only for ischemic stroke, NBP has been reported to increase the expression of N-methyl-D-aspartate subtype glutamate receptor 2B(NR2B) and synaptophysin in hippocampus of aged rats after chronic cerebral hypoperfusion and increasing brain acetylcholine level, which are important processes involved in learning and memory. It could alleviate the learning and memory deficits induced by cerebral ischemia in rats. A multicentre, randomized, double-blind, placebo-controlled trial conducted by Professor Jia investigated that NBP was effective for improving cognitive and global functioning in patients with subcortical vascular cognitive impairment without dementia and exhibited good safety over the 6-month treatment period. The pathogenesis of AD involved mitochondria dysfunction and microcirculation dysfunction, which are the action targets of NBP. Investigators observed that MMSE score lowering slowly when using NBP treatment in patients with mild to moderate AD already receiving donepezil. But investigators lack of system evaluation and follow-up. Hence, investigators hypothesized that NBP may have therapeutic efficacy for patients with AD and designed the present study.

ELIGIBILITY:
Inclusion Criteria:

* literate Chinese, aged 50-85 years, with a consistent caregiver who accompanied the subjects at least 4 days a week，2 hours a day;
* complaint and/or informant report of cognitive impairment involving memory and/or other cognitive domains lasting for at least 12 months; and progressing gradually.
* diagnosis of probable AD according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria;
* a mini-mental state examination (MMSE) score ≥11 and ≤22 (primary school) or ≥11 and ≤26 (junior school or above) ;
* Hachinski ischemia scale score ≤4;
* All patients meeting the clinical criteria underwent brain magnetic resonance imaging (MRI) scan including hippocampal assessment at screening. The MRI entry criteria are as follows: the number of cerebral infarcts (≥20 mm in diameter)less than 2, without infarcts in thalamus, hippocampal or entorhinal cortex, the medial temporal lobe atrophy visual rating scale (MTA) score more than 2 degree.
* absent of neurological sign;
* having used donepezil more than 3 months and remained relatively stable；
* sign the informed consent.

Exclusion Criteria:

* severe white matter lesion(WML)(score ≥3 according to the Fazekas rating scale), the number of cerebral infarcts (≥20 mm in diameter)more than 2, with infarcts in the important sites, such as thalamus, hippocampal or entorhinal cortex;
* dementia due to other causes, such as vascular dementia, infection of central nervous system，dementia with Lewy body(DLB)，etc
* suffered from other neurological disease, such as stroke, Parkinson's disease, epilepsy；
* suffered from mental disorders, such as schizophrenia，bipolar disorder，severe depression, delirium;
* suffered from unstable or severe disorders of heart, lung, liver, kidney and blood system;
* Severe impairment of vision and hearing;
* Using other cholinesterase inhibitors or memantine.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Mild to Moderate Alzheimer's Disease Already Receiving Donepezil
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Alzheimer's disease assessment scale-cognitive subscale (ADAS-cog) | Baseline, 48 weeks
  Primary efficacy parameter is the baseline- to-endpoint score change on ADAS-cog. The participants will be followed up every 12 weeks. There is five times interviews totally. The investigators compare the the baseline- to-endpoint score change on ADAS-cog at last.

SECONDARY OUTCOMES:
Clinician's Interview-Based Impression of Change Plus Caregiver Input (CIBIC-plus) | Baseline, 48 weeks
  secondary efficacy parameter is the endpoint score on CIBIC-plus
Alzheimer's Disease Cooperative Study-Activities of Daily Living(ADCS-ADL) | Baseline, 48 weeks
  Secondary efficacy parameter is the baseline-to-endpoint score change on the ADCS-ADL.The participants will be followed up every 12 weeks. There is five times interviews totally. The investigators compare the the baseline- to-endpoint score change on ADCS-ADL at last.
Neuropsychiatric Inventory(NPI) | Baseline, 48 weeks
  Additional parameter included the baseline-to-endpoint score changes on the NPI.The participants will be followed up every 12 weeks. There is five times interviews totally. The investigators compare the the baseline- to-endpoint score change on NPI at last.

CONTACTS AND LOCATIONS:
Overall Officials: qiu-min Qu, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes